CLINICAL TRIAL: NCT04418128
Title: Treatment Effect of Nafamostat Mesylate in Patients With COVID-19 Pneumonia: Open Labelled Randomized Controlled Clinical Trial
Brief Title: Clinical Efficacy of Nafamostat Mesylate for COVID-19 Pneumonia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, IN-GYU BAE, MD, Professor, Gyeongsang National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-04-012
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Corona Virus Infection; COVID-19
Keywords: Nafamostat; Pneumonia; TMPSS2; Serine protease inhibitor
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Pneumonia | interventions — nafamostat

STUDY DESIGN:
Intervention Model Description: This study is an open-labelled, randomized clinical trial to evaluate the efficacy of nafamostate in patients with COVID-19 pneumonia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (No Intervention): The conventional therapy comprised, as necessary, Lopinavir/ritonavir, Hydroxychlorquine, supplemental oxygen, Non-invasive and invasive ventilation, antibiotic agents, renal-replacement therapy (e.g.: CRRT, HD), extracorporeal membrane oxygenation (ECMO).
- Conventional therapy + Nafamostat mesylate (Experimental): * The conventional therapy comprised, as necessary, Lopinavir/ritonavir, Hydroxychlorquine, supplemental oxygen, Non-invasive and invasive ventilation, antibiotic agents, renal-replacement therapy (e.g.: CRRT, HD), extracorporeal membrane oxygenation (ECMO).
  * Nafamostat mesylate injection day), taking into account the severity and underlying disease of the clinical trial patient.
    * Method of administration: Nafamostat injection is mixed with 1,000 ml of 5% DW infusion, followed by continuous infusion over 24 hours.
    * Duration of administration: The researcher administers for 10-14 days considering the severity and underlying disease of the clinical trial patient.
  Interventions: Drug: Nafamostat Mesylate

INTERVENTIONS:
Drug: Nafamostat Mesylate — The Nafamostat mesilate group received continuous intravenous infusion of 0.1-0.2 mg/kg/h of nafamostat mesilate mixed with 5% DW.
  Arms: Conventional therapy + Nafamostat mesylate

SUMMARY:
In-vitro studies revealed that nafamostat mesylate has antiviral activity against Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and anti-inflammatory and anti-coagulation effect. However, there is no clinical studies on the efficacy of nafamostat in patients with COVID-19.

This study is conducted to evaluate the clinical efficacy of nafamostate mesylate in adult patients hospitalized with COVID-19 pneumonia.

DETAILED DESCRIPTION:
* The COVID-19 epidemic expanded to the whole world since it started from the Wuhan area in China in Dec. 2019. The Republic of Korea experiences a sharp increase in the patient since 24th Feb. 2020. An analysis of more than 70,000 patients in China, about 15% of them cause severe pneumonia, 5% require treatment in the intensive care unit, half of them die of the disease.
* There is no proven therapeutics for COVID-19 patients yet. Currently, the treatment with Kaletra, Hydroxychloroquine, etc. did not show apparent effect, and there are no other drugs that can apply to patients who get worse even with those drugs or severe.
* There are research reports that defective innate immunity and accelerated activation of the complement cascade, caused by the SARS-CoV-2, induce rapidly progressing pneumonitis.

  * Action mechanism of Nafamostat mesilate A. Show anti-viral effect by an inhibition serine protease, which is required for the host membrane fusion of viral envelop protein. In vitro experiments showed that the drug is effective in MERS-CoV, Influenza virus, and SARS-CoV-2.

B. Show anti-inflammatory effect by inhibition of the complement pathway, and inhibition of cytokine production.

This study is conducted to evaluate the clinical efficacy of nafamostate mesylate in adult patients hospitalized with COVID-19 pneumonia.

ELIGIBILITY:
* Inclusion Criteria:

  1. 18 years old or older
  2. Patients who have been confirmed of COVID-19 infection and has evidence for pneumonia

     * Confirmation of COVID-19 infection by RT-PCR of SARS-CoV-2
     * Definite diagnosis of new infiltration of the lungs by chest CT scan of chest radiographic inspection
  3. Patients who are within 72 hours of COVID-19 pneumonia confirmation
  4. Patients with 3(hospitalization, not requiring supplemental oxygen) or higher in seven-category ordinal scale of clinical status

     * Seven-category ordinal scale of clinical status

       1. not hospitalized with resumption of normal activities;
       2. not hospitalized, but unable to resume normal activities;
       3. hospitalization, not requiring supplemental oxygen;
       4. hospitalization, requiring supplemental oxygen;
       5. hospitalization, requiring nasal high-flow oxygen therapy and/or noninvasive mechanical ventilation;
       6. hospitalization, requiring extracorporeal membrane oxygenation and/or invasive mechanical ventilation;
       7. death.
  5. Patients who are eligible for diagnosis/evaluation to chest CT scan and related to it
  6. Patients should be able to understand the essence of the clinical trial and to submit a written consent document. For the patients who can understand the nature of the research but cannot sign the document, a relative can agree to the study.
* Exclusion Criteria:

  1. Patients who have a record of HIV or AIDS
  2. Female patients, either who are pregnant within 6 months before the investigation, who breast-fed babies within 3 months before the investigation, or who may get pregnant or breast-feed within 1 month after the investigation is over
  3. Patients at high risk of death within 3 days of randomized assignment, by the judge of the investigator
  4. Patients with liver cirrhosis whose Child-Puch score is B or C
  5. Patients who have liver disease abnormalities with ALT or AST > 5 times ULN
  6. Patients who can be in danger or who shows clinically-important other conditions which may interfere with the evaluation or completion of the test procedure, as the investigator's opinion
  7. Patients who are not appropriate for the test, as the investigator's opinion
  8. Patients who have hypersensitivity to the investigational drug

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-06-10 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with clinical improvement | Day 14 & Day 28
  Proportion of patients with clinical improvement as defined by live discharge from hospital or a decline of 2 categories on the seven-category ordinal scale of clinical status.
  * Seven-category ordinal scale of clinical status
  1. not hospitalized with resumption of normal activities;
  2. not hospitalized, but unable to resume normal activities;
  3. hospitalization, not requiring supplemental oxygen;
  4. hospitalization, requiring supplemental oxygen;
  5. hospitalization, requiring nasal high-flow oxygen therapy and/or noninvasive mechanical ventilation;
  6. hospitalization, requiring extracorporeal membrane oxygenation and/or invasive mechanical ventilation;
  7. death.

SECONDARY OUTCOMES:
Time to clinical improvement (TTCI) | up to 28 days
  Time to clinical improvement (TTCI) was defined as time from randomization to a decline of 2 categories on the seven-category ordinal scale of clinical status or live discharge from the hospital, whichever came first.
Clinical status assessed by 7-category ordinal scale | days 7, 14, and 28
  * Seven-category ordinal scale of clinical status
  1. not hospitalized with resumption of normal activities;
  2. not hospitalized, but unable to resume normal activities;
  3. hospitalization, not requiring supplemental oxygen;
  4. hospitalization, requiring supplemental oxygen;
  5. hospitalization, requiring nasal high-flow oxygen therapy and/or noninvasive mechanical ventilation;
  6. hospitalization, requiring extracorporeal membrane oxygenation and/or invasive mechanical ventilation;
  7. death.
     * Higher scores of Seven-category ordinal scale mean serious clinical status.
Change in National Early Warning Score (NEWS) | Day 1 trough Day 28
  The NEW score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness). The range of NEW score is from zero to 23. Higher scores of NEWS mean the higher risk of poor outcomes. The NEW Score is being used as an efficacy measure.
Time to National Early Warning Score (NEWS) of ≤ 2 and maintained for 24 hours | Day 1 through Day 28
Duration of hospitalization | Day 1 through Day 28
Duration of new non-invasive ventilation or high flow oxygen use | Day 1 through Day 28
Incidence of new non-invasive ventilation or high flow oxygen use | Day 1 through Day 28
Duration of new supplement oxygen use | Day 1 through Day 28
Incidence of new supplement oxygen use | Day 1 through Day 28
Duration of new ventilator or extracorporeal membrane oxygenation (ECMO) use | Day 1 through Day 28
Incidence of new ventilator or extracorporeal membrane oxygenation (ECMO) use | Day 1 through Day 28
Mortality at day 28 | Day 1 through Day 28
Time (days) from treatment initiation to death | Day 1 through Day 28
Proportions of patients with a negative nasopharyngeal swab and sputum sample for SARS-CoV-2 quantitative RT-PCR | days 3, 7, 10, 14, and 21
Viral load change (log10 viral load) of nasopharyngeal swab and sputum sample for SARS-CoV-2 quantitative RT-PCR | days 3, 7, 10, 14, and 21
Adverse events that occurred during treatment | Day 1 through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: IN-GYU BAE, MD, Principal Investigator — Gyeongsang National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gralinski LE, Sheahan TP, Morrison TE, Menachery VD, Jensen K, Leist SR, Whitmore A, Heise MT, Baric RS. Complement Activation Contributes to Severe Acute Respiratory Syndrome Coronavirus Pathogenesis. mBio. 2018 Oct 9;9(5):e01753-18. doi: 10.1128/mBio.01753-18. PMID 30301856
- [Background] Yamaya M, Shimotai Y, Hatachi Y, Lusamba Kalonji N, Tando Y, Kitajima Y, Matsuo K, Kubo H, Nagatomi R, Hongo S, Homma M, Nishimura H. The serine protease inhibitor camostat inhibits influenza virus replication and cytokine production in primary cultures of human tracheal epithelial cells. Pulm Pharmacol Ther. 2015 Aug;33:66-74. doi: 10.1016/j.pupt.2015.07.001. Epub 2015 Jul 10. PMID 26166259
- [Result] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Result] Hoffmann M, Schroeder S, Kleine-Weber H, Muller MA, Drosten C, Pohlmann S. Nafamostat Mesylate Blocks Activation of SARS-CoV-2: New Treatment Option for COVID-19. Antimicrob Agents Chemother. 2020 May 21;64(6):e00754-20. doi: 10.1128/AAC.00754-20. Print 2020 May 21. No abstract available. PMID 32312781
- [Derived] Moon K, Hong KW, Bae IG. Treatment effect of nafamostat mesylate in patients with COVID-19 pneumonia: study protocol for a randomized controlled trial. Trials. 2021 Nov 23;22(1):832. doi: 10.1186/s13063-021-05760-1. PMID 34814935